CLINICAL TRIAL: NCT06030882
Title: Improving Patient Outcomes Through the Implementation of a Standardized Biologic Care Pathway in the Treatment and Management of Inflammatory Bowel Disease Pathway in the Treatment and Management of Inflammatory Bowel Disease
Brief Title: Improving Patient Outcomes Through the Implementation of an IBD Biologic Care Pathway
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention (Biologic care pathway) was implemented outside of the context of a research study at our care centre, the QEII, as quality improvement. It became infeasible to consent all physicians to use the tool, and carry out this study.
Sponsor: Jennifer Jones (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Jennifer Jones, Gastroenterologist, Associate Professor, Department of Medicine, Dalhousie University, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 50757
Record Dates: First submitted 2023-07-10; First posted 2023-09-11 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: IBD; Biologics; Care Pathway
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biologic Care Pathway (Experimental): Care through a biologic care pathway
  Interventions: Other: Biologic Care Pathway
- Control (No Intervention): Care as usual

INTERVENTIONS:
Other: Biologic Care Pathway — Receiving care administered through a biologic care pathway.The central biologic intake nurse will touch base with the IBD program nurse navigator at preselected time points as per the pathway in order to coordinate the baseline pre- biologic work-up, clinical and biomarker assessments, and clinical assessments. Clinical management decisions will be informed by a combination of data points including clinical risk factors, TDM, fecal calprotectin concentrations, endoscopic and clinical disease activity indices as well as drug tolerance and adverse events. Within the care pathway, time- bound clinical and biomarker data will be provided to the treating clinician to help inform their clinical decisions.
  Arms: Biologic Care Pathway

SUMMARY:
Inflammatory Bowel Disease (IBD) includes a group of chronic inflammatory conditions of the gastrointestinal system and is composed of Crohn's disease and ulcerative colitis. As an immune-mediated disease, IBD treatment options include the use of biologic medicines including anti-tumor necrosis alpha factor (also called anti-TNFs) medication. Despite biologic medicines being an important part of IBD management, there is inconsistency in the way these medications are used. Implementation of evidence-based, standardized biologic care pathways (BCP) can improve treatment related outcomes. Previous research has shown that using a clinical care pathway, such as a BCP, is a feasible method to support clinical decision making and may improve disease-related outcomes for patients. The researchers propose a prospective study to determine how well a BCP can be incorporated into clinical practice, improve patient health outcomes, and reduce healthcare system redundancies. Also, the impact of a BCP on outcomes for patients treated with the help of a standardized BCP compared to those in patients treated without the use of a BCP will be studied. The results of this study will inform how best to incorporate evidence-based BCPs into real-world practice and support the wide-spread adoption of BCPs in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to age 18
* Starting an Anti TNF biologic therapy or Biosimilar

Exclusion Criteria:

* High-grade, symptomatic fibrostenotic strictures
* Perforating complications
* Intraabdominal or perianal abscesses
* Active infection,
* Known malignancy
* Any contraindication to biologic therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
EQ5D Score | week 0 (baseline)
  General Quality of life data measured using the Euroqol five dimension (EQ5D) Questionnaire. The EQ5D is a brief self-reported generic measure of current health. It is a 2 page questionnaire which has 5 descriptive questions. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
EQ5D Score | week 50
  General Quality of life data measured using the Euroqol five dimension (EQ5D) Questionnaire. The EQ5D is a brief self-reported generic measure of current health. It is a 2 page questionnaire which has 5 descriptive questions. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.

SECONDARY OUTCOMES:
Emergency room visits | week 0 (baseline)
  Number of emergency room visits
Emergency room visits | month 12
  Number of emergency room visits
inpatient hospitalization, | week 0
  Number of inpatient hospitalizations
inpatient hospitalization, | month 12
  Number of inpatient hospitalizations
disease-related surgery | week 0
  Number of disease related surgeries
disease-related surgery | month 12
  Number of disease related surgeries
ambulatory care visits | week 0
  number of ambulatory care visits
ambulatory care visits | month 12
  number of ambulatory care visits
drug therapy | week 0
  A list of current medications the patient is taking
drug therapy | month 12
  A list of current medications the patient is taking

OTHER OUTCOMES:
HBI Index Score | week 0 (baseline), week 12-14, week 30, week 50
  IBD disease activity measured by the Harvey Bradshaw Index (HBI index). The HBI involves patients answering five questions which are summed to produce a final score. The following are potential final score results:
  Remission: <5 Mild Disease: 5-7 Moderate Disease: 8-16 Severe Disease: >16
HBI Index Score | week 0 (baseline)
  IBD disease activity measured by the Harvey Bradshaw Index (HBI index). The HBI involves patients answering five questions which are summed to produce a final score. The following are potential final score results:
  Remission: <5 Mild Disease: 5-7 Moderate Disease: 8-16 Severe Disease: >16
HBI Index Score | week 12
  IBD disease activity measured by the Harvey Bradshaw Index (HBI index). The HBI involves patients answering five questions which are summed to produce a final score. The following are potential final score results:
  Remission: <5 Mild Disease: 5-7 Moderate Disease: 8-16 Severe Disease: >16
HBI Index Score | week 30
  IBD disease activity measured by the Harvey Bradshaw Index (HBI index). The HBI involves patients answering five questions which are summed to produce a final score. The following are potential final score results:
  Remission: <5 Mild Disease: 5-7 Moderate Disease: 8-16 Severe Disease: >16
HBI Index Score | week 50
  IBD disease activity measured by the Harvey Bradshaw Index (HBI index). The HBI involves patients answering five questions which are summed to produce a final score. The following are strata for final score results:
  Remission: <5 Mild Disease: 5-7 Moderate Disease: 8-16 Severe Disease: >16
Partial Mayo Score | week 0 (baseline)
  IBD disease activity (as measured by the Partial Mayo Score). Partial Mayo Score measures disease activity of Ulcerative colitis. The following are strata for final score results:
  Total Partial Mayo Index Score Remission: 0-1 Mild Disease: 2-4 Moderate Disease: 5-6 Severe Disease: 7-9
Partial Mayo Score | week 12
  IBD disease activity (as measured by the Partial Mayo Score). Partial Mayo Score measures disease activity of Ulcerative colitis. The following are strata for final score results:
  Total Partial Mayo Index Score Remission: 0-1 Mild Disease: 2-4 Moderate Disease: 5-6 Severe Disease: 7-9
Partial Mayo Score | week 30
  IBD disease activity (as measured by the Partial Mayo Score). Partial Mayo Score measures disease activity of Ulcerative colitis. The following are strata for final score results:
  Total Partial Mayo Index Score Remission: 0-1 Mild Disease: 2-4 Moderate Disease: 5-6 Severe Disease: 7-9
Partial Mayo Score | week 50
  IBD disease activity (as measured by the Partial Mayo Score). Partial Mayo Score measures disease activity of Ulcerative colitis. The following are strata for final score results:
  Total Partial Mayo Index Score Remission: 0-1 Mild Disease: 2-4 Moderate Disease: 5-6 Severe Disease: 7-9
Fecal calprotectin | week 0 (baseline)
  Fecal calprotectin concentration, assayed by stool sample
Fecal calprotectin | week 12
  Fecal calprotectin concentration, assayed by stool sample
Fecal calprotectin | week 30
  Fecal calprotectin concentration, assayed by stool sample
Fecal calprotectin | week 50
  Fecal calprotectin concentration, assayed by stool sample
CRP concentration | week 0 (baseline)
  serum CRP concentration
CRP concentration | week 12
  serum CRP concentration
CRP concentration | week 30
  serum CRP concentration
CRP concentration | week 50
  serum CRP concentration

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No